CLINICAL TRIAL: NCT00804531
Title: Intra-discal Steroid Injection for MODIC I Discopathy: A Randomized Control Trial
Brief Title: Intra-discal Steroid Injection for MODIC I Discopathy
Acronym: PREDID
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P070157
Record Dates: First submitted 2008-12-08; First posted 2008-12-09 (Estimated); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Back Pain Lower Back Chronic
Keywords: Low back pain; steroid injection; inter-vertebral disc; randomized trial; Lack of efficacy of usual recommended treatments; More than 40 on the pain numeric scale (0-100); Inflammatory discopathy (MODIC I) on MRI
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Visipaque - Hydrocortancyl (Experimental): Administration of two treatments for the experimental arm
  Interventions: Drug: Visipaque - Hydrocortancyl
- Visipaque (Placebo Comparator): Administration of only one treatment in intra discal of visipaque
  Interventions: Drug: Placebo comparator

INTERVENTIONS:
Drug: Visipaque - Hydrocortancyl — Visipaque 320 mg I/ml - 1 ml intra-discal route Hydrocortancyl 25 mg/ml - 1 ml intra-discal route
  Arms: Visipaque - Hydrocortancyl
Drug: Placebo comparator — Visipaque - 320 mg I/ml - 1 ml in intra-discal route
  Arms: Visipaque

SUMMARY:
To assess the efficacy on pain level at 1 month and 12 months of a steroid injection in the inter-vertebral disc for patients with chronic back pain and inflammatory discopathy on magnetic resonance imaging.

Hypothesis: delivering anti-inflammatory drugs in situ may decrease back pain in patients with inflammatory discopathy

DETAILED DESCRIPTION:
Objective: to assess the efficacy on pain level of a steroid injection in the inter-vertebral disc for patients with chronic back pain and MODIC I discopathy on MRI

Methods: a multicenter double blind randomized control trial Setting: 3 tertiary care hospitals in France Patients: 134 patients with disabling chronic low back pain not relieved by usual recommended treatments and MODIC I (inflammatory) discopathy on MRI Intervention: Injection of 25 mg of methylprednisolone in the inter-vertebral disc during a discography (intervention group, 67 patients) or discography alone (control group, 67 patients) Outcome measures: The primary outcome measure is pain level assessed on a 11-point numeric scale (0-100) at 1 month. Success is defined as less than 40 on pain numeric scale at 1 month. Secondary outcome measures are pain level at 12 months, Disability (Quebec questionnaire), quality of life (SF-12) at 1 and 12 months, anxiety and depression (HAD), analgesics and anti-inflammatories during the last week, return to work, assessment of the disabilities at 1 and 12 months and disc inflammation (on MRI) at 12 months. Tolerance and adverse effects will be recorded.

Trial duration: 36 months(24 months for inclusion and 12 months follow-up) Follow-up visits: at 1, 3, 6, and 12 months Statistical analysis: intention to treat

ELIGIBILITY:
Inclusion criteria :

* More than 18 and less than 70 years old
* Low back pain
* Daily pain for at least 3 months
* Pain level during the last 48 hours > 40 on the numeric pain scale (0-100)
* Lack of efficacy of usual recommended treatments and of other spine steroid injections (epidural or facet joints injections)
* Modic I discopathy on MRI
* Intra-discal injection at least 6 months before inclusion
* Written informed consent
* Social security
* Medical examination

Non inclusion criteria :

* Pregnancy
* Hypersensitivity to methylprednisolone or contrast
* Local or general infection
* Previous disc surgery less than 6 months
* Steroid treatment
* Previous infectious spondylodiscitis
* Ankylosing spondylitis
* Sciatica with neurologic defects
* Uncontrolled psychiatric conditions
* Inability to read or understand French language
* Anti-vitamin K treatments
* Severe coagulation diseases
* Fever > 38 or sedimentation rate > 20
* Discopathy with MODIC 1 signal on several different lumbar stages

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2009-04; Primary Completion 2015-05 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Back pain level assessed on a 11-point numeric scale (0-100) at 1 month. Success is defined as less than 40 on pain numeric scale at 1 month | 1 month

SECONDARY OUTCOMES:
pain level at 12 months | 12 months
Disability (Quebec questionnaire) | 1 month and 12 months
quality of life (SF-12) at 1 and 12 months | 1 month and 12 months
anxiety and depression (HAD) | 1 month and 12 months
disc inflammation (on MRI) at 12 month | 12 months
analgesics and anti-inflammatories during the last week | 1 month and 12 months
return to work | 1 month and 12 months
Assessment of the disabilities (scale of 6 classes) | 1 month and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Serge Poiraudeau, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Cochin, Paris, France

REFERENCES:
- [Background] Nguyen C, Boutron I, Baron G, Sanchez K, Palazzo C, Benchimol R, Paris G, James-Belin E, Lefevre-Colau MM, Beaudreuil J, Laredo JD, Bera-Louville A, Cotten A, Drape JL, Feydy A, Ravaud P, Rannou F, Poiraudeau S. Intradiscal Glucocorticoid Injection for Patients With Chronic Low Back Pain Associated With Active Discopathy: A Randomized Trial. Ann Intern Med. 2017 Apr 18;166(8):547-556. doi: 10.7326/M16-1700. Epub 2017 Mar 21. PMID 28319997
- [Derived] Daste C, Abdoul H, Foissac F, Lefevre-Colau MM, Poiraudeau S, Rannou F, Nguyen C. Patient acceptable symptom state for patient-reported outcomes in people with non-specific chronic low back pain. Ann Phys Rehabil Med. 2022 Jan;65(1):101451. doi: 10.1016/j.rehab.2020.10.005. Epub 2020 Nov 26. PMID 33152522